CLINICAL TRIAL: NCT00407576
Title: PET Imaging of Brain Amyloid Using [11C]MeS-IMPY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Robert B. Innis, M.D./National Institute of Mental Health, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 070036; 07-M-0036
Record Dates: First submitted 2006-12-02; First posted 2006-12-05 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-11-07

CONDITIONS: Alzheimer's Disease; Healthy
Keywords: Alzheimer's Disease; Positron Emission Tomography; Brain; Neurochemistry; Beta-Amyloid Plaques; PET; MeS-IMPY; Alzheimer Disease; AD; Dementia; Healthy Volunteer; HV
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — N,N-dimethyl-4-(6-(methylthio)imidazo(1,2-a)pyridine-2-yl)aniline

INTERVENTIONS:
Drug: [11C]MeS-IMPY

SUMMARY:
Alzheimer's disease is associated with accumulation in the brain of a protein called amyloid. The purpose of this study is to test the ability of a research drug to measure amyloid in brain using positron emission tomography (PET) and a research drug called [11C]MeS-IMPY.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is characterized pathologically by the presence of beta-amyloid plaques in brain. A substantial body of research indicates that the presence of increased beta -amyloid peptide is neurotoxic, and may initiate further pathology observed in AD including neurofibrillary tangles, synaptic loss and dysfunction, and neurodegeneration. There are multiple binding sites available on beta-amyloid plaques. Three clearly identified sites are Congo-red type, Thioflavin-T type, and FDDNP type. Radioligands currently under development using positron emission tomography (PET) for studying beta-amyloid in clinical research or drug development are based on Thioflavin-T site, such as [11C]PIB and [11C]SB-13. Though variously effective, these radioligands have one or more drawbacks with respect to measuring relative regional beta-amyloid densities. Therefore, we have recently developed [11C]MeS-IMPY as an alternative radioligand for imaging beta-amyloid, which will allow a more accurate quantification of amyloid plaques in AD brain. In the current protocol, we wish to evaluate [11C]MeS-IMPY in both healthy subjects and AD patients to determine the kinetics of brain imaging beta-amyloid plaques in AD patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy control subjects aged 18-90 years and AD patients aged 50-90, with history/physical exam, ECG, and laboratory tests.

Informed Consent.

AD Patients: Mini-Mental State Examination (score greater than or equal to 10).

AD Patients: Meet NINCDS-ADRDA criteria for probable AD.

EXCLUSION CRITERIA:

1. Current or prior history of any alcohol or drug abuse.
2. Severe systemic disease based on history and physical exam.
3. Positive result on urine screen for illicit drugs.
4. Laboratory tests with clinically significant abnormalities.
5. Prior participation in other research protocols or clinical care in the last year such that radiation exposure would exceed the annual limits.
6. Pregnancy or breast feeding.
7. Claustrophobia.
8. Presence of ferromagnetic metal in the body or heart pacemaker.
9. History of brain disease other than Alzheimer's disease.
10. Unable to lay on one's back for the PET/MRI scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-12-01; Primary Completion 2008-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Agdeppa ED, Kepe V, Liu J, Flores-Torres S, Satyamurthy N, Petric A, Cole GM, Small GW, Huang SC, Barrio JR. Binding characteristics of radiofluorinated 6-dialkylamino-2-naphthylethylidene derivatives as positron emission tomography imaging probes for beta-amyloid plaques in Alzheimer's disease. J Neurosci. 2001 Dec 15;21(24):RC189. doi: 10.1523/JNEUROSCI.21-24-j0004.2001. PMID 11734604
- [Background] Burger C, Buck A. Requirements and implementation of a flexible kinetic modeling tool. J Nucl Med. 1997 Nov;38(11):1818-23. PMID 9374364
- [Background] Ichise M, Toyama H, Innis RB, Carson RE. Strategies to improve neuroreceptor parameter estimation by linear regression analysis. J Cereb Blood Flow Metab. 2002 Oct;22(10):1271-81. doi: 10.1097/01.WCB.0000038000.34930.4E. PMID 12368666